CLINICAL TRIAL: NCT05210218
Title: Effect on Weight Loss of an Oral Association of Cinnamon Bark (Cinnamomum Cassia) and Withania Somnifera in Adult Patients With Overweight or Obesity: a Randomized, Prospective, Placebo-controlled, Multicenter, Cross-over, Pilot Study
Brief Title: Cinnamon and Withania on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Full Professor MD PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE5115
Record Dates: First submitted 2021-12-29; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mildly hypocaloric diet + CC 300 mg +WS 150 mg tid (Experimental): The study product, in a capsule formulation, was made by the extract of Cinnamomum cassia (CC) and Withania somnifera (WS) (300 mg+150mg, respectively) (Nutrintech Ltd., London, UK) to be taken three times a day. All patients received a mildly hypocaloric diet (i.e., -20% of the usual caloric intake as assessed by a 24-hour dietary recall).
  Interventions: Dietary Supplement: Cinnamomum cassia (CC) and Withania somnifera (WS) (300 mg+150mg, respectively)
- mildly hypocaloric diet + placebo tid (Placebo Comparator): Each patient took the placebo (i.e., the same amount of cellulose). All patients received a mildly hypocaloric diet (i.e., -20% of the usual caloric intake as assessed by a 24-hour dietary recall).
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Cinnamomum cassia (CC) and Withania somnifera (WS) (300 mg+150mg, respectively) — The study product, in a capsule formulation, was made by the extract of Cinnamomum cassia (CC) and Withania somnifera (WS) (300 mg+150mg, respectively) (Nutrintech Ltd., London, UK)
  Arms: mildly hypocaloric diet + CC 300 mg +WS 150 mg tid
Dietary Supplement: placebo — cellulose
  Arms: mildly hypocaloric diet + placebo tid

SUMMARY:
With the prevalence of obesity soaring and the absence of an effective and safe treatment that is low-cost and always feasible, the use of food supplements has gained attention for the potential benefits in the absence of significant safety concerns. Cinnamon (CC) and Withania somnifera (WS) are plant-based supplements reported to be effective in improving metabolic health and body composition, the first mainly acting on insulin resistance and the second on energy expenditure and leptin resistance, as shown in preclinical and some clinical studies. Their association, possibly synergistic leveraging different mechanisms of action, has never been studied.

This was a double-blind placebo-controlled study. Patients with overweight or obesity were prescribed a mildly hypocaloric diet with CC 300 mg plus WS 150 mg tid for 4 weeks in a cross over design and anthropometric parameters together with safety outcomes were collected.

ELIGIBILITY:
Inclusion Criteria:

* age range: 25-75 years
* overweight or obesity (BMI range: 26-35)

Exclusion Criteria:

* heart failure
* congenital cardiomyopathies
* episodes of tachy/brady-arrythmias
* acute myocardial infarction within 3 months from the enrollment
* inability or unwillingness to provide informed consent
* pregnancy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
weight change | at baseline and at every follow up visit, through study completion, an average of 10 weeks
  body mass change in kg

SECONDARY OUTCOMES:
waist circumference change | at baseline and at every follow up visit through study completion, an average of 10 weeks
  waist circumference change in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request to the corresponding author